CLINICAL TRIAL: NCT05444738
Title: Efficacy of Administering Oxytocin Orally Using a Medicated Lollipop Approach on Peripheral Concentrations and Attention: Comparisons With Intranasal and Lingual Spray Administration
Brief Title: Effects of Oxytocin Administered Orally Using a Medicated Lollipop on Peripheral Concentrations and Attention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Principal Inverstigator, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-86
Record Dates: First submitted 2022-06-20; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: social salience; oral oxytocin; antisaccade paradigm; attention
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled triple-blind between-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral oxytocin (Experimental): oral lollipop with oxytocin (24IU)
  Interventions: Drug: oral lollipop with oxytocin (24IU)
- oral lollipop with placebo (Placebo Comparator): Placebo orally (identical ingredients, except the active agent)
  Interventions: Drug: oral lollipop with placebo

INTERVENTIONS:
Drug: oral lollipop with oxytocin (24IU) — Immediately before drug administration, a blood sample (5ml) is collected. For drug administration, participants will be instructed to suck the lollipop medicated with 24IU oxytocin for 3 minutes and then to sit relaxed in a quiet room for 30 minutes prior to taking another blood sample (5ml). Participants then start the anti-saccade attention task 45 minutes after drug administration.
  Other Names: oral oxytocin
  Arms: oral oxytocin
Drug: oral lollipop with placebo — Immediately before drug administration, a blood sample (5ml) is collected. For placebo administration, participants will be instructed to suck the placebo lollipop for 3 minutes and then to sit relaxed in a quiet room for 30 minutes prior to taking another blood sample (5ml). Participants then start the anti-saccade attention task 45 minutes after placebo administration.
  Other Names: oral placebo
  Arms: oral lollipop with placebo

SUMMARY:
The study will investigate whether oxytocin (24IU) administered orally using medicated lollipops results in increased peripheral oxytocin concentrations and can modulate social attention in an anti-saccade paradigm in the same way as when it is administered by intranasal or lingual routes.

DETAILED DESCRIPTION:
In a triple-blind, placebo-controlled experiment, 72 adult male subjects will be randomly allocated to either receive oral oxytocin (24IU - medicated lollipop - n = 36) or placebo (lollipop without oxytocin - n = 36). After treatment allocation, all subjects will first fill out a set of questionnaires as a control for potential confounders, including Beck Depression Inventory-II (BDI), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), the Second Version of Social Responsiveness Scale (SRS-2), Childhood Trauma Questionnaire (CTQ), Toronto Alexithymia Scale (TAS), and Positive Affect Negative Affect Scale (PANAS). Immediately before and 30 minutes after oral treatment administration, subjects will have 5 ml blood samples taken for assay of oxytocin concentrations. Subjects will sit quietly and relax in between blood samples. After the second blood sample, subjects will be positioned sitting in front of an eye-tracking machine and briefly practicing the anti-saccade task. Subjects will then perform the full anti-saccade eye-tracking task, which includes both social (emotional faces - angry, fear, happy, sad, and neutral) and non-social (oval shapes or houses) stimuli (similar to previous studies using intranasal -see NCT03486925 and NCT04493515). After the task, subjects will be asked to guess which treatment they received, and their ability to do so analyzed using chi-squared. Treatment effects on primary (anti-saccade and pro-saccade errors and response latencies) outcomes will be analyzed using ANOVAs. In a secondary analysis, associations between primary outcome measures and basal and altered oxytocin concentrations will be analyzed using Pearson or Spearman correlations. Additionally, a comparison between the effects of oxytocin administered intranasally, lingually (using previously published data), and orally (medicated lollipop) on outcome measures will be analyzed using ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

1. History of brain injury
2. Head trauma
3. Substance abuse
4. Medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Oral oxytocin effect on error rates of saccade/anti-saccade to social (faces) and non-social (shape) cues between the oxytocin and placebo groups. | 45minutes ~ 100 minutes after oral lollipop
  A mixed ANOVA to compare differences in error rates in saccade/anti-saccade to different conditions (social/non-social) between two treatment groups.
Oral oxytocin effect on latencies (in milliseconds) of saccade/anti-saccade to social (faces) and non-social (shape) cues between the oxytocin and placebo groups. | 45minutes ~ 100 minutes after oral lollipop
  A mixed ANOVA to compare differences of latencies (in milliseconds) in saccade/anti-saccade to different conditions (social/non-social) between two treatment groups.

SECONDARY OUTCOMES:
Plasma oxytocin concentrations (pg/ml) before (basal) and 30 minutes after oral oxytocin or placebo administration. | 30 minutes after oral lollipop
  Differences in plasma oxytocin concentrations between the two treatment groups before and after the oral administration will be analyzed using mixed ANOVA, with time point and treatment group as independent variables.
Change of Mood as assessed by the Positive Affect Negative Affect Scale (PANAS) before and after the experiment in two treatment groups. | 45minutes ~ 100 minutes after oral lollipop
  The Positive Affect Negative Affect Scale (PANAS) measures both positive and negative emotions in a person. The Positive Affect score range from 10-50, with higher scores representing higher levels of positive affect. The Negative Affect scores range from 10-50, with lower scores representing lower levels of negative affect.
  The differences in PANAS scores in pre-/post-experiment between treatment groups will be analyzed using mixed ANOVA.
Change of state anxiety as assessed by the State-Trait Anxiety Inventory (STAI) before and after the experiment in two treatment groups. | 45minutes ~ 100 minutes after oral lollipop
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of the trait (TAI) and state (SAI) anxiety. Each type of anxiety has its own scale of 20 different questions that are scored, and scores range from 20-80, with higher scores indicating greater anxiety.
  Differences in state anxiety (SAI) scores in pre-/post-experiment between treatment groups will be analyzed using mixed ANOVA.
Associations between plasma oxytocin concentration changes and task performance (error rates, latencies), mood (PANAS), and state anxiety (SAI). | 45minutes ~ 100 minutes after oral lollipop
  Pearson or Spearman correlation analysis between plasma oxytocin concentration changes (%) and error rates (%).
  Pearson or Spearman correlation analysis between plasma oxytocin concentration changes (%) and latencies in milliseconds.
  Pearson or Spearman correlation analysis between plasma oxytocin concentration changes (%) and post-task PANAS scores.
  Pearson or Spearman correlation analysis between plasma oxytocin concentration changes (%) and post-task SAI scores.
Comparison between the effects of oxytocin administered intranasally, lingually, and orally on anti-saccade errors (%) by mixed ANOVA. | 45minutes ~ 100 minutes after oral lollipop
  Comparisons between anti-saccade errors in the current oral oxytocin administration experiment and those in previous ones using intranasal and lingual oxytocin administration (NCT03486925 and NCT04493515) will be made using mixed ANOVAs, with route (intranasal/lingual/oral) and treatment (oxytocin/placebo) as between-subject factors, condition (social/non-social) as within-subject factor.
Comparison between the effects of oxytocin administered intranasally, lingually, and orally on latencies in milliseconds by mixed ANOVA. | 45minutes ~ 100 minutes after oral lollipop
  Comparisons between anti-saccade latencies (in milliseconds) in the current oral oxytocin administration experiment and those in previous ones using intranasal and lingual oxytocin administration (NCT03486925 and NCT04493515) will be made using mixed ANOVAs, with route (intranasal/lingual/oral) and treatment (oxytocin/placebo) as between-subject factors, condition (social/non-social) as within-subject factor.
Comparison between the effects of oxytocin administered intranasally, lingually, and orally in state anxiety (measured by the State-Trait Anxiety Inventory) changes by mixed ANOVA. | 45minutes ~ 100 minutes after oral lollipop
  The State-Trait Anxiety Inventory (STAI) measures both trait (TAI) and state (SAI) anxiety. Each type of anxiety has its own scale of 20 different questions that are scored, and scores range from 20-80, with higher scores indicating greater anxiety.
  Comparisons between changes of state anxiety (SAI) in the current oral oxytocin administration experiment and those in previous ones using intranasal and lingual oxytocin administration (NCT03486925 and NCT04493515) will be made using mixed ANOVAs, with route (intranasal/lingual/oral) and treatment (oxytocin/placebo) as between-subject factors, condition (social/non-social) as within-subject factor.
  changes = (post-task SAI scores - pre-task SAI scores).

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technolog, Chengdu, Sichuan, China

REFERENCES:
- [Background] Xu X, Li J, Chen Z, Kendrick KM, Becker B. Oxytocin reduces top-down control of attention by increasing bottom-up attention allocation to social but not non-social stimuli - A randomized controlled trial. Psychoneuroendocrinology. 2019 Oct;108:62-69. doi: 10.1016/j.psyneuen.2019.06.004. Epub 2019 Jun 15. PMID 31229634
- [Background] Zhuang Q, Zheng X, Yao S, Zhao W, Becker B, Xu X, Kendrick KM. Oral Administration of Oxytocin, Like Intranasal Administration, Decreases Top-Down Social Attention. Int J Neuropsychopharmacol. 2022 Nov 17;25(11):912-923. doi: 10.1093/ijnp/pyac059. PMID 36053298